CLINICAL TRIAL: NCT03842423
Title: Brachial Plexus Block in Children and Adolescents Requiring Surgery Following Trauma
Brief Title: Brachial Plexus Block in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Haider, Principal Investigator, Medical University of Vienna
Other Study IDs: 2090/2018
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Upper Extremity Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: All patients under the age of 18 who were treated for upper extremity injuries between 2002 and 2018 and receiving brachial plexus anaesthesia.
  Interventions: Procedure: Brachial Plexus Anaesthesia

INTERVENTIONS:
Procedure: Brachial Plexus Anaesthesia — Regional anaesthesia for treatment of upper extremity injuries.

SUMMARY:
This study involves a retrospective evaluation of brachial plexus anaesthesia in children and adolescents (patients under the age of 18) undergoing surgical procedures of the upper extremity following trauma. The investigators plan to recruit patients from our hospital patient database meeting our inclusion criteria. Observational period was defined between 1st of January 2002 and 31st of October 2018. Necessity to convert to general anaesthesia was defined as primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Brachial plexus anaesthesia for surgical intervention of upper extremity injuries

Exclusion Criteria:

* age above 18

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under the age of 18 who sustained an injury of the upper extremity requiring surgery and received brachial plexus anaesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 2760 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Conversion to general anaesthesia | intraoperatively
  The necessity to convert to general anaesthesia will be obtained from surgery and anaesthesiology protocols and serves as primary outcome to evaluate efficacy of the investigated method of anaesthesia. All patients who received plexus brachialis anaesthesia but had to be converted to general anaesthesia during or prior the surgical intervention will assigned to this outcome measurement. Number of patients who required conversion will be given as percentage of total patient collective. Possible variables: e.g. 0=no conversion, 1=conversion.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zadrazil M, Opfermann P, Marhofer P, Westerlund AI, Haider T. Brachial plexus block with ultrasound guidance for upper-limb trauma surgery in children: a retrospective cohort study of 565 cases. Br J Anaesth. 2020 Jul;125(1):104-109. doi: 10.1016/j.bja.2020.03.012. Epub 2020 Apr 24. PMID 32340734